CLINICAL TRIAL: NCT05125393
Title: Evaluation the Safety of Indocyanine Green Guided Treatment of Henle Trunk Using Endoscopic Linear Stapler in Laparoscopic Radial Hemicolectomy of Colon Cancer -- a Prospective Randomized Controlled Multicenter Clinical Study (SIGHELC)
Brief Title: Evaluation the Safety of Indocyanine Green Guided Treatment of Henle Trunk
Acronym: SIGHELC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai East Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Shanghaieasthospital-2021216
Record Dates: First submitted 2021-09-13; First posted 2021-11-18 (Actual); Last update posted 2021-11-18 (Actual); Status verified 2021-11

CONDITIONS: Colon Cancer; Surgery
Keywords: Colon cancer; Henle trunk; Linear stapler; Laparoscopic surgery
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Linear stapler group (Experimental): In the experimental group, indocyanine green was injected for development during the operation after ileocolic vessel and the middle colonic vessel were dissected. The tributary vessels of the Henle trunk were disconnected with a linear stapler if there was no obvious lymph node development, which means ligated not in the root. Otherwise, they were transferred to the experimental group.
  Interventions: Procedure: Laparoscopic linear stapler
- Conventional group (No Intervention): The branches of Henle trunk were dissected according to the conventional method and clamped at the root.

INTERVENTIONS:
Procedure: Laparoscopic linear stapler — The ileocecal or ascending colon tumors were resected using a combined cephalic caudal approach. When the accessory right colonic vein is separated from the head and then turned to the caudal side for upward dissociation. After no metastasis of 203 groups of lymph nodes is confirmed according to ICG development during the operation, the Henle stem and its root tissue were resected with a linear stapler.
  Arms: Linear stapler group

SUMMARY:
Laparoscopic right hemicolectomy D3 dissection or complete mesocolic excision (CME) has become the standard treatment for right hemi-colon cancer, and the treatment of Henle trunk is one of the difficulties of the operation. However, there are many variations in the Henle trunk, and the vein wall is thin. It is very easy to damage the Henle trunk and its branches during the operation, resulting in massive bleeding, especially for beginners. In addition, retrospective studies found that for ileocecal or ascending colon tumors, low ligation of Henle trunk can obtain better lymph node clearance. In the early stage, the investigators improved the surgical method for ileocecal or ascending colon tumors. An endoscopic linear stapler was used to disconnect the surrounding tissues of Henle trunk under the guidance of indocyanine green developer. The retrospective study of small samples found that it can significantly reduce the incidence of local bleeding, shorten the operation time, and obtain the same lymph node clearance rate. At present, there is less large-scale randomized controlled study on the disconnection of Henle trunk with linear stapler for right colon cancer. In recent years, the were nearly 1000 cases/year of colorectal cancer operated in department of gastrointestinal surgery of shanghai east hospital. Therefore, the investigators plan to cooperate with many domestic colorectal cancer treatment centers to take the lead in carrying out this prospective, multicenter and randomized controlled trail, to explore the safety and efficacy of linear stapler in the treatment of Henle trunk in laparoscopic radial hemicolectomy of colon cancer. The investigators hope to provide accurate clinical evidence for individualized precision treatment of rectal cancer patients.

DETAILED DESCRIPTION:
Laparoscopic right hemicolectomy D3 dissection or complete mesocolic excision (CME) has become the standard treatment for right hemi-colon cancer, and the treatment of Henle's trunk is one of the difficulties of the operation. The traditional view is that D3 lymph node dissection should be performed routinely in the right hemicolectomy, that is, the blood vessels of the right hemi-colon including the Henle trunk and its tributary should be ligated at the level of superior mesenteric artery and vein, and the lymph nodes should be cleaned. However, there is a large degree of variation in the anatomy of Henle trunk, which is even considered as the "fingerprint" of CME in the right colon. Coupled with the thin venous wall, it is very easy to damage Henle trunk and its branches during operation and resulting in massive bleeding, especially for beginners. In addition, a retrospective study found that the lymph node metastasis rate around the middle colonic vein and Henle trunk was less than 5% in ileocecal or ascending colon tumors. Low ligation in this area can also obtain a better lymph node resection rate.

Based on the above points, the investigators propose to improve the surgical method in ileocecal or ascending colon tumors using a combined cephalic caudal approach. When the accessory right colonic vein is separated from the head and then turned to the caudal side for upward dissociation. After no metastasis of 203 groups of lymph nodes is confirmed according to indocyanine green (ICG) development during the operation, the Henle trunk and its root tissue were resected with a linear stapler. The investigators believe that this method has the following advantages: 1. The Henle trunk together with the branches could be effectively disconnect, which can reduce the difficulty of operation and shorten the learning curve; 2. The incidence of bleeding was reduced. Our preliminary small sample studies have confirmed that the improved operation does not increase postoperative complications and can obtain the same oncological prognosis.

This is a prospective, multicenter, randomized, parallel controlled trial designed to evaluate the safety and efficacy of linear stapler in laparoscopic radical resection of ascending colon cancer. The total number of patients enrolled in this study is 128, including 64 in the control group and 64 in the experimental group. In the experimental group, indocyanine green was injected for development during the operation after ileocolic vessel and the middle colonic vessel were dissected. The tributary vessels of the Henle trunk were disconnected with a linear stapler if there was no obvious lymph node development, which means ligated not in the root. Otherwise, they were transferred to the experimental group. In the control group, the branches of Henle's trunk were dissected according to the conventional method and clamped at the root. The main research objectives include: 1. Intraoperative bleeding volume 2. Operation time. Secondary research objectives included: 1. Lymph node detection rate 2. R0 resection rate 3. Complication rate 4. At least one serious complication rate within 30 days after resection.

At present, there is less large-scale randomized controlled study on the disconnection of Henle trunk with linear stapler for right colon cancer. In recent years, the were nearly 1000 cases/year of colorectal cancer operated in department of gastrointestinal surgery of shanghai east hospital. Therefore, the investigators plan to cooperate with many domestic colorectal cancer treatment centers to take the lead in carrying out this prospective, multicenter and randomized controlled trail, to explore the safety and efficacy of linear stapler in the treatment of Henle trunk in laparoscopic radial hemicolectomy of colon cancer. The investigators hope to provide accurate clinical evidence for individualized precision treatment of rectal cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with locally advanced colorectal cancer met the following criteria at the time of enrollment:

  1. Adult male and female, aged between 18-75 years
  2. Colonoscopic biopsy confirmed colonic adenocarcinoma
  3. Before treatment, the tumor was located between ileocecal part and ascending colon liver area
  4. There were no local complications (no complete obstruction, no massive active bleeding, no perforation and abscess formation) before operation
  5. The functions of heart, lung, liver and kidney meet the requirements of operation and anesthesia
  6. Informed consent form be signed

Exclusion Criteria:

* Patients who met the following criteria at the time of inclusion were excluded from this trial:

  1. Previous history of malignant colorectal tumor
  2. Patients with intestinal obstruction, intestinal perforation and intestinal bleeding requiring emergency surgery
  3. The primary tumor invades the abdominal wall and / or adjacent organs, resulting in inability to R0 resection
  4. Unresectable lymph node metastasis
  5. Recent diagnosis complicated with other malignant tumors
  6. Patients who had participated or were participating in other clinical trials within 4 weeks before enrollment
  7. American Society of Anesthesiologists (ASA) physical status classes ≥ grade IV and / or Eastern Cooperative Oncology Group (ECOG) physical state score ≥ 2 points (see Appendix for details)
  8. Patients with severe liver and kidney function, cardiopulmonary function, coagulation dysfunction or combined with serious basic diseases can not tolerate the operation
  9. Have a history of serious mental illness
  10. Pregnant or lactating women
  11. Patients with uncontrolled infection before operation
  12. Some researchers believe that patients with other clinical and laboratory conditions should not participate in the trial

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2021-12-01 (Estimated); Primary Completion 2023-12-01 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Intraoperative bleeding | From the beginning to the end of the operation
  The total amount of bleeding during the operation, that is, the total amount of blood loss in the drainage bottle and gauze
Operation time | From the beginning to the end of the operation
  Time from start to end of operation

SECONDARY OUTCOMES:
Number of lymph nodes dissected | 7 days after operation
  Number of lymph nodes dissected
R0 resection rate | 7 days after operation
  Percentage of patients with R0 resection
Incidence of complications | within 30 days after resection
  Percentage of postoperative complications
Incidence of at least one serious complication within 30 days after resection | within 30 days after resection
  Incidence of at least one serious complication within 30 days after resection，such as Massive hemorrhage, anastomotic fistula, septic shock, death, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaohua Jiang, Doctor, Study Chair — Shanghai East Hospital